CLINICAL TRIAL: NCT01678950
Title: Comparison Between MostCare and Echo-Doppler for Cardiac Output Measurement: an Observational Study
Brief Title: MostCare Versus Echo-Doppler for Cardiac Output Measurement
Acronym: PRAM
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Responsible Party: Principal Investigator, Sabino Scolletta, MD, Principal Investigator, Azienda Ospedaliera Universitaria Senese
Other Study IDs: PRAM2012
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Cardiac Output Measurement
Keywords: Cardiac output monitoring; Echocardiography; Pulse contour system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Recently, an uncalibrated minimally invasive Pulse-code Modulator (PCM) has been developed: the MostCare system. This monitoring system is powered by Pressure Recording Analytical Method (PRAM), which is based on the mathematical analysis of the arterial pressure profile changes. It allows beat-to-beat Stroke Volume (SV) assessment from the pressure signal recorded invasively in radial, brachial, or femoral arteries. The most innovative features of this method are: 1) the lack of a calibration requirement, 2) the analysis of the arterial wave signal is performed at 1000 Hz, 3) a dedicated arterial catheter-transducer is unnecessary. MostCare is powered by PRAM (Pressure Recording Analytical Method) algorithm. The investigators primary end-point was to evaluate the relationship between Cardiac Output (CO) measured by MostCare with CO calculated with Echo-Doppler in Intensive Care Unit (ICU) patients under different clinical conditions. As a secondary end-point the investigators evaluated the relationship between CO measured by MostCare with CO obtained with thermodilution techniques (standard bolus thermodilution or transpulmonary thermodilution, i.e. PiCCO system). This is a prospective multicentre observational study.

DETAILED DESCRIPTION:
(*) Study design

A. MostCare system data acquisition Before each CO measurement, the arterial pressure catheter and transducer quality will be assessed as follows: easy aspiration of 5 ml of blood easily re-injected without resistance; visual assessment of the quality of the arterial waveform contour; adequate response to the flush test (square wave). If necessary, the best position for the signal quality will be checked by extending the wrist and manipulating the catheter. For each determination of Echo-Doppler (and ThD-CO when applicable), a corresponding value for MostCare must be obtained by averaging the individual beats over the same time necessary to obtain the Echo-doppler-CO (and ThD-CO when applicable) measurements.

B. Echo-Doppler data acquisition (transoesophageal - TOE - or transthoracic - TTE - echo) Echo-Doppler-CO will be measured using the standard formula CSA x VTI (cross sectional area x velocity time integral x heart rate in ml/min). 2D measurement of the aortic annulus diameter allows calculation of the flow CSA which is then multiplied by the VTI (velocity time integral) of the Pulsed Doppler flow velocity profile across the aortic valve to determine the SV.

Other hemodynamic variables as an ancillary part of the study will compare shortening fraction (SF) or EF fraction from Echocardiography with CCE and dp/dt.

C. Thermodilution data acquisition (ThD-CO) (when applicable) Data coming from ThD pulmonary artery catheter (PAC) or a CVC + femoral artery catheter (transpulmonary thermodilution, PiCCO system) will be collected from the monitor itself or the system for patient monitoring used in the units.

For standard PAC-ThD-CO, five consecutive injections of 10 ml of 5% glucose cold solution will be randomly injected during respiratory cycle over a 5-min period. Thermodilution-CO (or PiCCO-CO) will be calculated as the average of the five measurements. All these 5 measurements will be collected.

MostCare, Echo-doppler (and Thermodilution when applicable) Change in ventilator parameters, sedation drugs, or fluid infusions or vasopressor dose will not be allowed during the acquisition time.

(*) Study timing and procedure

For each patient CO determinations will be performed as follows:

Mandatory measurements:

• Baseline: (MostCare + Echo-doppler simultaneously, and MostCare + Echo-doppler + Thermodilution when applicable) = single comparison between techniques.

Recorded but not mandatory measurements (fitting to the therapeutic protocol used in each center):

• Pre- and post- treatment (fluid challenge, vasoactive drugs and inotropics changes) (MostCare + Echo-doppler simultaneously, and MostCare + Echo-doppler + Thermodilution when applicable) = dynamic comparison between techniques (two measures). This will allow a sub-analysis of CO (the trend of CO) changes, validity of trend, for both SV and CO before and after a therapeutic intervention.

Data to be collected:

Patient: demographic, anthropometric, pre-medical history, indication(s) for ICU admission; (cardiovascular diseases and cardiac function, respiratory diseases, etc...), severity scores (SAPS II, SOFA, ….).

All patients enrolled will be analysed in intention-to-treat even data recording failed. In this case, that would be a limit if any, for the tested technique.

Hemodynamic MostCare: SV, HR, CO, CCE, ∆P/∆T, ABPs, ABPd, ABPm. Other hemodynamic data: CVP, PaoP, SvO2, lactate,... Echocardiography: stroke volume, heart rate, cardiac output. Other hemodynamic variables are allowed to be collected by Echo according to the centre protocols and the experience of each centre.

Cardiac and vasoactive drugs dose or infusion rate will be collected: dobutamine, dopamine, norepinephrine, epinephrine, nitrates, beta-blockers, ACE-I,ecc.

Ventilatory: mechanical ventilation settings: mode of ventilation (CPAP, BiPAP, VC, PC), pressure support (if applicable), peak and plateau pressure, PEEP level, FiO2 oxygenation (SaO2, PaO2,…) ICU stay and outcome: morbidity (number and type of complications), length of stay, mortality.

(*) Statistical analysis and methodology, number of patients to be enrolled, duration of the study:

Collected data will be copied on an excel file to be properly independently analyzed with a statistical software. Correlation tests (Spearman or Pearson), Student paired t-test, and Bland-Altman analysis will be applied. A minimum of 30 patients per centre will be enrolled in the study in a period of 18 months.

This "minimum number" of patients is mandatory as: 1) the enrollment of 30 patients per centre eliminates the potential bias that may occur when few data come from a single centre, 2) minimum 300 patients enrolled represents a suitable number to obtain the "statistical power" necessary to validate the comparison between the different methods, and 3) further analysis and comparisons in subgroup of patients having similar clinical settings can be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients equipped with a standard arterial catheter-line (femoral or radial artery) for invasive arterial blood pressure monitoring.
* Patients requiring an echocardiographic evaluation - Transthoracic Echocardiographic Evaluation (TEE)or Transesophageal Echocardiographic Evaluation (TOE) - as a routine need or in the context of Acute Cardiocirculatory failure with suspected implication of cardiac dysfunction or Acute Respiratory failure and suspicion of cardiac failure.
* *When a pulmonary artery catheter (PAC, standard bolus thermodilution, ThD) is used or a central venous catheter linked with a femoral artery catheter to measure the transpulmonary thermodilution (PiCCO system: Continuous pulse contour cardiac analysis), the comparison will be done as a secondary end point of the protocol.

  * The point n.3 is optional

Exclusion Criteria:

* Related to MostCare:

pathologies that could affect the quality and reliability of the arterial signal (aortic valve pathologies, aortic aneurysms) and arrhythmias that generate hemodynamic instability (i.e., variations in mean BP measurements > 10%); poor quality of the arterial pressure signal after a standard flush test (i.e., over-damped or under-damped arterial trace).

* Related to Echo-Doppler: non-feasibility to obtain a fulfilled quality of the images.
* Patients younger than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Intensive Care Unit, under different clinical conditions
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
cardiac output | comparison of monitoring systems
  comparison of cardiac output monitoring systems

CONTACTS AND LOCATIONS:
Locations (14):
- Department of Anesthesiology & Intensive Care - Lariboisière University Hospital University Paris 7 Diderot. France, Paris, Paris, France
- Italy (11):
  - Department of Anaesthesia and Intensive Care, Torrette University Hospital, Ancona, Ancona
  - Intensive Care Unit, Santa Maria Annunziata Hospital, Florence, Florence
  - Department of Cardiovascular Anesthesia and Intensive Care, Careggi University Hospital, Italy, Florence, Florence
  - Anaesthesia and Intensive Care Unit, S. Giovanni di Dio - Torregalli Hospital, Florence, Florence
  - Department of Anaesthesia and Intensive Care, Ospedali Riuniti Foggia University Hospital, Foggia, Foggia
  - Cardio-Thoracic-Vascular Anaesthesia and Intensive Care, San Raffaele University Hospital, Milan, Milan
  - Department of Anaesthesia and Intensive Care, Pisa University Hospital, Pisa, Pisa
  - Cardiovascular Anesthesia, Policlinico Umberto I°, Rome, Rome
  - Department of Anaesthesia and Intensive Care, Siena University Hospital, Siena, Siena
  - Policlinico Universitario Padova, Padua
  - Ospedale S. Antonio Abate di Pontremoli, Pontremoli
- of Anesthesia, Critical Care and Pain Medicine, Hospital Universitario de la Ribera, Valencia, Valencia, Spain
- (Cardiothoracic Anaesthesia, Heart and Lung Centre, New Cross Hospital, Wolverhampton, England, United Kingdom